CLINICAL TRIAL: NCT06046157
Title: Effect of Oral Motor Intervention on Feeding Parameters in Preterm Babies
Brief Title: Oral Motor Intervention for Preterm Babies
Acronym: PIOMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc İlknur Budancamanak (Unknown); Professor Kadir Şerafettin Tekgündüz (Unknown); Associate Professor Mustafa Kara (Unknown); MSc Ebru Betül Albayrak (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Director, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B. 30.2. ATA.0.01.00/702
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Preterm Babies
Keywords: Premature infant oral motor intervention (PIOMI); Premature; Nutrition
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast milk-scented PIOMI (Experimental): During PIOMI application, the baby will be smelled his/her own breast milk.
  Interventions: Other: Breast milk-scented PIOMI
- Breast milk-tasting PIOMI (Experimental): During PIOMI application, the baby will be able to taste his own breast milk. The finger on which PIOMI was applied will be immersed in breast milk.
  Interventions: Other: Breast milk-tasting PIOMI
- Control (No Intervention): Only PIOMI application will be made.

INTERVENTIONS:
Other: Breast milk-scented PIOMI — During PIOMI, the scent of breast milk will be provided through cotton soaked in breast milk placed 1.5 cm away from the babies.
  PIOMI: Oral motor intervention for premature infants is a standardized oral motor therapy for preterm infants that has been shown to have strong intervention fidelity and has been tested internationally.
  It is a 5-minute, 8-step focused therapy designed to help the premature baby respond functionally to lip, chin and lip movements and pressure, applied for 7 consecutive days using all aseptic precautions with gloved fingers.
  Intervention provides assisted movement to activate muscle contraction and movement against resistance to build strength.
  Arms: Breast milk-scented PIOMI
Other: Breast milk-tasting PIOMI — The finger used during PIOMI application will be performed by dipping it into breast milk. This will ensure that babies taste breast milk.
  PIOMI: Oral motor intervention for premature infants is a standardized oral motor therapy for preterm infants that has been shown to have strong intervention fidelity and has been tested internationally.
  It is a 5-minute, 8-step focused therapy designed to help the premature baby respond functionally to lip, chin and lip movements and pressure, applied for 7 consecutive days using all aseptic precautions with gloved fingers.
  Intervention provides assisted movement to activate muscle contraction and movement against resistance to build strength.
  Arms: Breast milk-tasting PIOMI

SUMMARY:
The goal of this clinical trial is to evaluate the effect of oral motor intervention (PIOMI) applied to preterm babies along with the smell and taste of breast milk on feeding parameters and the transition time to oral feeding. The main questions it aims to answer are:

* Does affect nutritional parameters PIOMI with the smell of breast milk?
* Does affect nutritional parameters PIOMI with breast milk taste? Participants will consist of breast milk-scented PIOMI, breast milk-tasting PIOMI and control groups.

Researchers will compare breast milk-scented PIOMI, breast milk-tasting PIOMI and control groups to see if early feeding skills.

DETAILED DESCRIPTION:
The preterm newborn population is potentially unable to be fed orally for a long time during the postnatal period. Since the physiological functions of preterm babies have not yet matured, their adaptation to the external uterine environment is more complicated. This also means long hospital stays for premature babies. One of the main criteria for a preterm baby to be discharged from the hospital is to be able to feed orally.

Premature oral motor intervention (PIOMI) is included in the literature as one of the treatment programs to improve the oral motor control and neurobehavioral status of preterm babies. No study design has been found regarding PIOMI, which is applied to preterm babies with the smell and taste of breast milk. This research was planned to evaluate the effect of oral motor intervention (PIOMI) applied to preterm babies along with the smell and taste of breast milk on feeding parameters.

ELIGIBILITY:
Inclusion Criteria:

* Breastfed,
* Preterm babies with a gestational age of 28-32 weeks,
* No facial deformity,
* No respiratory, cardiovascular, gastrointestinal or neurological disorders or syndromes that would prevent or complicate oral feeding,
* It will produce preterm babies who are not fed orally but are fed via tube (orogastric).

Exclusion Criteria:

* Having respiratory distress,
* Babies who do not receive informed consent form from the parents will not be included.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Early feeding skills | 12 week
  EFS was revised to evaluate the feeding skills of preterm infants. The EFS 19 items in 5 subscales: respiratory regulation, oral-motor function, swallowing coordination, engagement, and physiologic stability.
  The tool includes items that evaluate the development of oral feeding skills and items that describe observable indicators of a problem during feeding. Items related to feeding skills are evaluated using the following 3-option structure: skill not yet observed 1, skill emerging 2 and skill consistently observed 3 with minor variations in wording depending on the item. Indicators of problems within a skill are scored using a frequency-based 3-option structure: frequent indication of problem 1, occasional indication of problem 2, and never or rare indication of a problem 3 and again, the specific wording varies by item. The overall EFS score is the sum of the 5 subscale scores and ranges from 19 to 57. Higher scores indicate more mature feeding skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No